CLINICAL TRIAL: NCT00280605
Title: Study of the Outcome of Patients With Lower Urinary Symptoms Suggestive of Benign Prostatic Hyperplasia and Treated With Alfuzosin 10 mg Once Daily for 3 Months in China
Brief Title: ALF-ONE : ALFuzosin ONcE Daily
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0168
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

INTERVENTIONS:
Drug: Alfuzosin

SUMMARY:
The aim of the study is to collect, under daily practice conditions, clinical data on the safety profile and the efficacy of a new formulation of alfuzosin administered once daily in patients with lower urinary tract symptoms (LUTS) suggestive of benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients suffering from Lower Urinary Tract Symptoms suggestive of Benign Prostatic Hyperplasia

Exclusion Criteria:

* Patients requiring Benign Prostatic Hyperplasia surgery immediately or within the 12 following months
* Patients previously not improved by an alpha 1-blocker treatment
* Patients whose urinary symptoms are satisfactorily controlled on other Benign Prostatic Hyperplasia medication (alpha 1-blockers and 5-ARI)
* Known hypersensitivity to alfuzosin
* History of postural hypotension or syncope
* Combination with other alpha 1-blockers
* Hepatic insufficiency
* Unstable angina pectoris
* Severe concomitant condition threatening life

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2005-08; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Spontaneous adverse events
Blood pressure and heart rate measured in sitting position
International Prostate Symptom Score (IPSS) and quality of life index
DAN-PSS sexual function score
PSA levels measured at baseline
Maximum flow rate and residual urine

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Blayney, MD, Study Director — Sanofi